CLINICAL TRIAL: NCT02475850
Title: Randomized Trial of a Multifactorial Fall Injury Prevention Strategy
Brief Title: Strategies to Reduce Injuries and Develop Confidence in Elders
Acronym: STRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Yale University (Other); University of California, Los Angeles (Other); Healthcare Partners (Other); The University of Texas Medical Branch, Galveston (Other); University of Pittsburgh Medical Center (Other); Johns Hopkins University (Other); Sinai Health System (Other); Reliant Medical Group (Other); Partners HealthCare (Other); University of Michigan (Other); University of Iowa (Other); Essentia Health (Other); Wake Forest University (Other); National Institute on Aging (NIA) (NIH); Patient-Centered Outcomes Research Institute (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy Latham, Study Director, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U01AG048270 (NIH); 1U01AG048270-01 (NIH)
Record Dates: First submitted 2015-06-01; First posted 2015-06-19 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Accidental Falls; Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fall prevention standard of care (Other): An evidence-based patient-centered intervention that will combine elements of a multifactorial, risk factor-based, standardly-tailored fall prevention strategy developed at Yale, practice guidelines offered by the CDC's "STEADI" toolbox and the joint American Geriatrics Society/British Geriatrics Society guidelines, and ACOVE practice change approach
  Interventions: Other: Evidence-based tailored fall prevention
- Control (Other): Usual fall prevention care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Evidence-based tailored fall prevention
  Arms: Fall prevention standard of care
Other: Usual care
  Arms: Control

SUMMARY:
The aim of this pragmatic cluster-randomized trial is to determine the effectiveness of an evidence-based, patient-centered multifactorial fall injury prevention strategy in community dwelling older adults at risk of falls recruited from 86 primary care practices around the U.S.

DETAILED DESCRIPTION:
Objective: To determine the effectiveness of an evidence-based, patient-centered multifactorial fall injury prevention strategy implemented within primary care practices using usual health care resources

Design: This study is a cluster randomized, parallel group superiority trial with practices stratified by healthcare system and patients nested within practices. The unit of randomization is the practice.

Study Duration: The total study duration is 5 years. Recruitment will take place over 20 months, with follow-up taking place for 24 months - 44 months depending on date of enrollment.

Trial Sites: 86 primary care practices that are part of 10 trial sites located around the U.S.: The Partners' Health Care System; Essentia; Hopkins Health Care System; HealthCare Partners; Reliant Health Care System; Mount Sinai Health Care System; University of Pittsburgh Health Care System; University of Texas Medical Branch Health Care System; University of Iowa Health Care System; University of Michigan Health Care System.

Number of Subjects: The original target sample size was 6,000 participants enrolled in 86 practices to provide 90% power to detect a 20% reduction in the rate of the primary outcome with intervention relative to control. The study was originally designed for a study duration of 36 months with 18 months of recruitment and a minimum of 18 months of follow-up. The study was extended to a 44 month study (20 months of recruitment and a minimum 24 month of follow-up). For a 44 month trial, it was estimated that a sample size of 5,322 subjects would provide 90% power to detect a 20% reduction in the rate of the primary outcome with the intervention relative to control.

Main Inclusion Criteria Community-living persons, 70 years or older, who are at increased risk for serious fall injuries.

Intervention: An evidence-based patient-centered intervention that will combine elements of a multifactorial, risk factor-based, standardly-tailored fall prevention strategy developed at Yale, practice guidelines offered by the Center for Disease Control's (CDC's) "STEADI" toolbox (Stopping Elderly Accidents, Disability and Injury) and the joint American Geriatrics Society/British Geriatrics Society guidelines, and Assessing Care of Vulnerable Elders (ACOVE) practice change approach. The fall prevention strategies will be systematically implemented into clinical practice using: delivery system design to improve quality (Co-management); decision support (algorithms); information systems (software); self-management support (patient/caregiver engagement and activation); and linkage to community-based resources.

Primary Outcome: The primary outcome is adjudicated serious fall injuries, operationalized as a fall resulting in: (1) (fracture other than thoracic/lumbar vertebral; joint dislocation; or cut requiring closure) AND any medical attention; OR (2) (head injury; sprain or strain; bruising or swelling; or other) requiring hospitalization.

Primary Analysis: The risk of any serious fall injury (i.e., time to first event) will be analyzed using a survival model that incorporates competing risks (due to death) and clustering. In this analysis, participants who are lost to follow-up without a prior serious fall-related injury will be censored at their date last seen. In a sensitivity analysis, the investigators will adjust for the pre-specified set of baseline covariates to examine their influence on the intervention effect.

Secondary Outcomes: All self-reported falls, all self-reported fall-related injuries, and measures of well-being.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 70 years of age.
* The patient must answer 'yes' to one or more of the following questions:
* Have you fallen and hurt yourself in the past year?
* Have you fallen 2 or more times in the past year?
* Are you afraid that you might fall because of balance or walking problems?

Exclusion Criteria:

* The patient is enrolled in hospice.
* The patient resides in a nursing home.
* The patient is not capable of providing informed consent (or assent), and a proxy is not available.
* The patient does not speak English or Spanish

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5451 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital; Thomas Gill, MD, Principal Investigator — Yale University; Dave Reuben, MD, Principal Investigator — University of California, Los Angeles; Nancy Latham, PhD, Study Director — Brigham and Women's Hosptial
Locations (10):
- United States (10):
  - Healthcare Partners, Torrance, California
  - University of Iowa Health Alliance, Des Moines, Iowa
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Partners Healthcare, Boston, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - Mt Sinai Health System, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch at Galveston, Galveston, Texas

REFERENCES:
- [Derived] Esserman D, Greene EJ, Latham NK, Kane M, Lu C, Peduzzi PN, Gill TM, Ganz DA. Assessing readiness to use electronic health record data for outcome ascertainment in clinical trials - A case study. Contemp Clin Trials. 2024 Jul;142:107572. doi: 10.1016/j.cct.2024.107572. Epub 2024 May 11. PMID 38740298
- [Derived] Ganz DA, Gill TM, Reuben DB, Bhasin S, Latham NK, Peduzzi P, Greene EJ. Costs of fall injuries in the STRIDE study: an economic evaluation of healthcare system heterogeneity and heterogeneity of treatment effect. Cost Eff Resour Alloc. 2023 Aug 2;21(1):49. doi: 10.1186/s12962-023-00459-3. PMID 37533073
- [Derived] Ganz DA, Yuan AH, Greene EJ, Latham NK, Araujo K, Siu AL, Magaziner J, Gurwitz JH, Wu AW, Alexander NB, Wallace RB, Greenspan SL, Rich J, Volpi E, Waring SC, Dykes PC, Ko F, Resnick NM, McMahon SK, Basaria S, Wang R, Lu C, Esserman D, Dziura J, Miller ME, Travison TG, Peduzzi P, Bhasin S, Reuben DB, Gill TM. Effect of the STRIDE fall injury prevention intervention on falls, fall injuries, and health-related quality of life. J Am Geriatr Soc. 2022 Nov;70(11):3221-3229. doi: 10.1111/jgs.17964. Epub 2022 Aug 6. PMID 35932279
- [Derived] Esserman DA, Gill TM, Miller ME, Greene EJ, Dziura JD, Travison TG, Meng C, Peduzzi PN. A case study of ascertainment bias for the primary outcome in the Strategies to Reduce Injuries and Develop Confidence in Elders (STRIDE) trial. Clin Trials. 2021 Apr;18(2):207-214. doi: 10.1177/1740774520980070. Epub 2021 Mar 7. PMID 33678038
- [Derived] Gill TM, Bhasin S, Reuben DB, Latham NK, Araujo K, Ganz DA, Boult C, Wu AW, Magaziner J, Alexander N, Wallace RB, Miller ME, Travison TG, Greenspan SL, Gurwitz JH, Rich J, Volpi E, Waring SC, Manini TM, Min LC, Teresi J, Dykes PC, McMahon S, McGloin JM, Skokos EA, Charpentier P, Basaria S, Duncan PW, Storer TW, Gazarian P, Allore HG, Dziura J, Esserman D, Carnie MB, Hanson C, Ko F, Resnick NM, Wiggins J, Lu C, Meng C, Goehring L, Fagan M, Correa-de-Araujo R, Casteel C, Peduzzi P, Greene EJ. Effect of a Multifactorial Fall Injury Prevention Intervention on Patient Well-Being: The STRIDE Study. J Am Geriatr Soc. 2021 Jan;69(1):173-179. doi: 10.1111/jgs.16854. Epub 2020 Oct 9. PMID 33037632
- [Derived] Bhasin S, Gill TM, Reuben DB, Latham NK, Ganz DA, Greene EJ, Dziura J, Basaria S, Gurwitz JH, Dykes PC, McMahon S, Storer TW, Gazarian P, Miller ME, Travison TG, Esserman D, Carnie MB, Goehring L, Fagan M, Greenspan SL, Alexander N, Wiggins J, Ko F, Siu AL, Volpi E, Wu AW, Rich J, Waring SC, Wallace RB, Casteel C, Resnick NM, Magaziner J, Charpentier P, Lu C, Araujo K, Rajeevan H, Meng C, Allore H, Brawley BF, Eder R, McGloin JM, Skokos EA, Duncan PW, Baker D, Boult C, Correa-de-Araujo R, Peduzzi P; STRIDE Trial Investigators. A Randomized Trial of a Multifactorial Strategy to Prevent Serious Fall Injuries. N Engl J Med. 2020 Jul 9;383(2):129-140. doi: 10.1056/NEJMoa2002183. PMID 32640131
- [Derived] Esserman D. From screening to ascertainment of the primary outcome using electronic health records: Challenges in the STRIDE trial. Clin Trials. 2020 Aug;17(4):346-350. doi: 10.1177/1740774520920898. Epub 2020 May 14. PMID 32408769
- [Derived] Gill TM, McGloin JM, Shelton A, Bianco LM, Skokos EA, Latham NK, Ganz DA, Nyquist LV, Wallace RB, Carnie MB, Dykes PC, Goehring LA, Doyle M, Charpentier PA, Greene EJ, Araujo KL. Optimizing Retention in a Pragmatic Trial of Community-Living Older Persons: The STRIDE Study. J Am Geriatr Soc. 2020 Jun;68(6):1242-1249. doi: 10.1111/jgs.16356. Epub 2020 Mar 25. PMID 32212395
- [Derived] Ganz DA, Siu AL, Magaziner J, Latham NK, Travison TG, Lorenze NP, Lu C, Wang R, Greene EJ, Stowe CL, Harvin LN, Araujo KLB, Gurwitz JH, Agrawal Y, Correa-De-Araujo R, Peduzzi P, Gill TM; STRIDE Investigators. Protocol for serious fall injury adjudication in the Strategies to Reduce Injuries and Develop Confidence in Elders (STRIDE) study. Inj Epidemiol. 2019 Apr 15;6:14. doi: 10.1186/s40621-019-0190-2. eCollection 2019. PMID 31245263
- [Derived] Gill TM, McGloin JM, Latham NK, Charpentier PA, Araujo KL, Skokos EA, Lu C, Shelton A, Bhasin S, Bianco LM, Carnie MB, Covinsky KE, Dykes P, Esserman DA, Ganz DA, Gurwitz JH, Hanson C, Nyquist LV, Reuben DB, Wallace RB, Greene EJ. Screening, Recruitment, and Baseline Characteristics for the Strategies to Reduce Injuries and Develop Confidence in Elders (STRIDE) Study. J Gerontol A Biol Sci Med Sci. 2018 Oct 8;73(11):1495-1501. doi: 10.1093/gerona/gly076. PMID 30020415

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Fall Prevention Standard of Care: An evidence-based patient-centered intervention that will combine elements of a multifactorial, risk factor-based, standardly-tailored fall prevention strategy developed at Yale, practice guidelines offered by the CDC's "STEADI" toolbox and the joint American Geriatrics Society/British Geriatrics Society guidelines, and ACOVE practice change approach
  Evidence-based tailored fall prevention
- Control: Usual fall prevention care
  Usual care
Period: Overall Study
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Started | 2802 | 2649
Completed | 2209 | 2165
Not Completed | 593 | 484
Not completed — Death | 155 | 141
Not completed — Lost to Follow-up | 217 | 188
Not completed — Withdrawal by Subject | 221 | 155

BASELINE CHARACTERISTICS:
Groups:
- Intervention: An evidence-based patient-centered intervention that will combine elements of a multifactorial, risk factor-based, standardly-tailored fall prevention strategy developed at Yale, practice guidelines offered by the CDC's "STEADI" toolbox and the joint American Geriatrics Society/British Geriatrics Society guidelines, and ACOVE practice change approach
  Evidence-based tailored fall prevention
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 2649 | 2802 | 5451
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.5 (5.8) | 79.9 (5.7) | 79.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1629 | 1752 | 3381
  Male | 1020 | 1050 | 2070
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 211 | 196 | 407
  Not Hispanic or Latino | 2428 | 2592 | 5020
  Unknown or Not Reported | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 26 | 44 | 70
  Native Hawaiian or Other Pacific Islander | 1 | 5 | 6
  Black or African American | 164 | 128 | 292
  White | 2394 | 2571 | 4965
  More than one race | 22 | 16 | 38
  Unknown or Not Reported | 38 | 34 | 72
Positive on Fall Risk Screening Questions [Count of Participants; unit: Participants]
  Fallen 2 or more times in past year | 896 | 1015 | 1911
  Fallen and hurt yourself in past year | 1031 | 1089 | 2120
  Fear of falling because of balance or walking problems | 2274 | 2405 | 4679
Educational Level [Count of Participants; unit: Participants]
  High school graduate or less | 643 | 602 | 1245
  Some college or equivalent | 659 | 697 | 1356
  College graduate or higher | 1343 | 1502 | 2845
  Unknown | 4 | 1 | 5
Chronic coexisting conditions - number per participant [Mean (Standard Deviation); unit: number chronic conditions per subject] | 2.1 (1.3) | 2.1 (1.3) | 2.1 (1.3)
Clinically significant cognitive impairment [Count of Participants; unit: Participants] — Four or more errors on 6-item Callahan cognitive screener OR the interview was completed entirely by proxy
  Participants | 75 | 85 | 160
Use of mobility aid or inability to ambulate [Count of Participants; unit: Participants] | 909 | 972 | 1881
Number of positive responses to screening questions regarding fall injuries [Count of Participants; unit: Participants]
  1 | 1571 | 1634 | 3205
  2 | 605 | 629 | 1234
  3 | 473 | 539 | 1012
History of fracture other than of the hip after 50 yr of age [Count of Participants; unit: Participants] | 876 | 918 | 1794
History of hip fracture after 50 years of age [Count of Participants; unit: Participants] | 119 | 132 | 251

OUTCOME MEASURES:

1. Primary Outcome: First Adjudicated Serious Fall-Related Injury
Description: Number of first adjudicated serious fall-related injury serious fall-related injury events per 100 per years of follow-up.
Time Frame: Enrollment through last completed follow-up or death interview (max 44 months)
Measure: Number (95% Confidence Interval); unit: events per 100 person years of follow-up
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 2802 | 2649
events per 100 person years of follow-up | 4.87 [4.31 to 5.43] | 5.34 [4.55 to 6.13]
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.245, Regression, Cox — p<0.05 threshold (primary outcome); multistate model accounting for death as a semi-competing risk; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.80 to 1.06]

2. Secondary Outcome: First Self-reported Fall-related Injury
Description: Number of first self-reported fall-related injuries per 100 per years of follow-up
Time Frame: Enrollment through last completed follow-up or death interview (max 44 months)
Measure: Number (99% Confidence Interval); unit: events per 100 person years of follow-up
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 2802 | 2649
events per 100 person years of follow-up | 25.64 [24.19 to 27.08] | 28.62 [26.53 to 30.72]
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.004, Regression, Cox — p< 0.01 threshold (secondary outcome); Hazard Ratio (HR) = 0.90, 99% CI 2-sided [0.83 to 0.99]

3. Secondary Outcome: Time to Self-reported Falls
Description: ** data for this outcome was not collected
Time Frame: these data were not collected
Population: These data were not collected
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Physical Function
Description: Late Life Function and Disability Instrument (LL-FDI) function score. The scores are on a 0-100 scale, higher score = better function. The measure reported is the mean of scores at the 12-month and 24-months follow-up assessment
Time Frame: measured at 12-month and 24-month follow-up assessments, reported score is an average (mean) of the follow-up scores
Population: subsample selected for well-being measures with completed baseline LL-FDI
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 380 | 358
units on a scale | 58.45 (0.48) | 57.73 (0.51)
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.309, Mixed Models Analysis — p < 0.01 threshold (secondary outcome); random: patients nested within practices; fixed: baseline score, randomization constraint vars, predictors of missingness; Difference in least-squared means across = 0.72, 99% CI 2-sided [-1.10 to 2.54], Standard Error of Mean 0.71

5. Secondary Outcome: Disability
Description: Late Life Function and Disability Instrument (LL-FDI) disability score. The scores are on a 0-100 scale, higher score = less disability. The measure reported is the mean of scores at the 12-month and 24-months follow-up assessment
Time Frame: measured at 12-month and 24-month follow-up assessments, reported score is an average (mean) of the follow-up scores
Population: subsample selected for well-being measures with completed baseline LL-FDI
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 380 | 358
units on a scale | 55.16 (0.63) | 54.57 (0.67)
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.528, Mixed Models Analysis — p < 0.01 threshold (secondary outcome); [statistical method as in outcome 4, analysis 1]; Least squares means = 0.59, 99% CI 2-sided [-1.80 to 0.93]

6. Secondary Outcome: Anxiety
Description: Patient-reported Outcome Measure Information System (PROMIS) Anxiety subscale. Measured on a 8-40 Scale, higher score = more anxiety.
Time Frame: Measured at 12-month and 24-month follow-up assessments, reported score is an average (mean) of the follow-up scores.
Population: subsample selected for well-being measures and with completed baseline PROMIS Anxiety
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Fall Prevention Standard of Care: An evidence-based patient-centered intervention that will combine elements of a multifactorial, risk factor-based, standardly-tailored fall prevention strategy developed at Yale, practice guidelines offered by the CDC's "STEADI" toolbox and the joint American Geriatrics Society/British Geriatrics Society guidelines, and ACOVE practice change approach
  Evidence-based tailored fall prevention
Arm/Group | Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 371 | 350
units on a scale | 11.63 (0.29) | 12.53 (0.30)
Statistical Analysis 1: Comparison: Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.037, Mixed Models Analysis — p < 0.01 threshold (secondary outcome); [statistical method as in outcome 4, analysis 1]; Least squares means = -0.90, 99% CI 2-sided [-2.00 to 0.20], Standard Error of Mean 0.43 — Difference in least-squared means across all follow-up (repeated measures: 12 months/24 months)

7. Secondary Outcome: Depression
Description: PROMIS depression subscale. Measured on a 8-40 Scale, higher score = more depression.
Time Frame: Measured at 12-month and 24-month follow-up assessments, reported score is an average (mean) of the follow-up scores.
Population: subsample selected for well-being measures and with completed baseline PROMIS dep
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 372 | 350
units on a scale | 11.75 (0.31) | 12.94 (0.32)
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.009, Mixed Models Analysis — p<0.01 threshold (secondary outcome); [statistical method as in outcome 4, analysis 1]; Least squares means = -1.19, 99% CI 2-sided [-2.36 to -0.02], Standard Error of Mean 0.45

8. Secondary Outcome: Fear of Falling
Description: Falls Efficacy Scale. Measured on a 10-40 Scale, higher score = more fear of falling.
Time Frame: Measured at 12-month and 24-month follow-up assessments, reported score is an average (mean) of the follow-up scores.
Population: subsample selected for well-being measures and with completed baseline FES
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
Number analyzed (Participants) | 372 | 351
units on a scale | 16.03 (0.35) | 16.10 (0.37)
Statistical Analysis 1: Comparison: Intervention - Fall Prevention Standard of Care vs Control; Test type: Superiority; p = 0.897, Mixed Models Analysis — p <0.01 threshold (secondary outcome); [statistical method as in outcome 4, analysis 1]; Least squares means = -0.07, 99% CI 2-sided [-1.38 to 1.25], Standard Error of Mean 0.51 — Difference in least-squared means across all follow-up (repeated measures: 12 months, 24 months)

ADVERSE EVENTS:
Time Frame: Enrollment through death, withdrawal, or end of study (max 44 months)
Description: Only SAEs (death and hospitalization) were recorded. AEs were not collected in this pragmatic trial.
Arm/Group | Intervention - Fall Prevention Standard of Care | Control
All-Cause Mortality (participants affected / at risk) | 235/2802 | 220/2649
Serious Adverse Events (participants affected / at risk) | 1139/2802 | 1108/2649
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention - Fall Prevention Standard of Care (N=2802) | Control (N=2649)
hospitalization (Blood and lymphatic system disorders) | 24 (29) | 29 (34)
hospitalization (Cardiac disorders) | 199 (270) | 199 (259)
hospitalization (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
hospitalization (Ear and labyrinth disorders) | 7 (7) | 3 (3)
hospitalization (Endocrine disorders) | 7 (7) | 7 (8)
hospitalization (Eye disorders) | 4 (4) | 5 (5)
hospitalization (Gastrointestinal disorders) | 161 (208) | 135 (176)
hospitalization (General disorders) | 159 (194) | 152 (168)
hospitalization (Hepatobiliary disorders) | 11 (13) | 17 (19)
hospitalization (Immune system disorders) | 4 (4) | 1 (1)
hospitalization (Infections and infestations) | 252 (324) | 231 (298)
hospitalization (Injury, poisoning and procedural complications) | 187 (225) | 196 (242)
hospitalization (Investigations) | 21 (22) | 32 (35)
hospitalization (Metabolism and nutrition disorders) | 54 (59) | 55 (70)
hospitalization (Musculoskeletal and connective tissue disorders) | 173 (205) | 156 (182)
hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 (59) | 52 (58)
hospitalization (Nervous system disorders) | 178 (230) | 153 (192)
hospitalization (Psychiatric disorders) | 26 (31) | 24 (30)
hospitalization (Renal and urinary disorders) | 51 (54) | 55 (67)
hospitalization (Reproductive system and breast disorders) | 8 (8) | 6 (6)
hospitalization (Respiratory, thoracic and mediastinal disorders) | 156 (196) | 119 (156)
hospitalization (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (6)
hospitalization (Social circumstances) | 5 (6) | 2 (2)
hospitalization (Vascular disorders) | 101 (116) | 119 (135)
hospitalization (Vascular disorders) | 63 (72) | 77 (91)
hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT02475850/SAP_000.pdf
  • Study Protocol (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT02475850/Prot_001.pdf